CLINICAL TRIAL: NCT00107783
Title: Long-Term Clinical Trial of Nitisinone in Alkaptonuria
Brief Title: Long-Term Study of Nitisinone to Treat Alkaptonuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: William A. Gahl, M.D./National Human Genome Research Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 050076; 05-HG-0076 (Other: NHGRI)
Record Dates: First submitted 2005-04-07; First posted 2005-04-08 (Estimated); Results first posted 2011-01-19 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2010-12

CONDITIONS: Alkaptonuria
Keywords: Arthritis; Homogentisic Acid; Corneal Damage; Tyrosine; Alkaptonuria; Photophobia; Nitisinone
MeSH Terms: conditions — Alkaptonuria; Arthritis; Corneal Injuries; Photophobia | interventions — nitisinone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): No treatment
- Nitisinone-treated (Experimental): Subjects received nitisinone 2 mg orally, once daily.
  Interventions: Drug: Nitisinone (NTBC)

INTERVENTIONS:
Drug: Nitisinone (NTBC) — Treatment
  Other Names: Orfadin
  Arms: Nitisinone-treated

SUMMARY:
This 3-year study will examine the safety and effectiveness of long-term use of nitisinone (Orfadin) for treating joint problems in patients with alkaptonuria, an inherited disease in which a compound called homogentisic acid accumulates. The excess homogentisic acid causes arthritis and limited joint movement. It can also cause heart valve damage and kidney stones.

Patients between 30 and 80 years of age with alkaptonuria may be eligible for this study. Patients must have hip involvement, but at least one remaining hip joint. Candidates are recruited from among patients enrolled in protocol 00-HG-0141, "Clinical, Biochemical, and Molecular Investigations into Alkaptonuria." Participants may enter both protocols simultaneously.

Participants are randomly assigned to one of two treatment groups: one group takes their regular medicines plus a 2-mg nitisinone capsule daily; the other group takes only their regular medicines. Patients taking nitisinone have blood tests to measure liver function 2 weeks and 6 weeks after starting treatment. Before starting therapy, all patients are admitted to the NIH Clinical Center for 4-5 days to undergo the following procedures:

* Medical history and physical examination
* 24-hour urine collection to test for sugar, protein, and other molecules
* Blood tests for liver and thyroid function, blood counts, and blood chemistries
* Blood and urine tests to measure tyrosine and other amino acids and homogentisic acid
* Bone x-rays
* Spiral CT (computed tomography) of the abdomen to detect kidney stones
* Eye examination and evaluations by specialists in rehabilitation medicine and pain, plus other consults in skin, brain, lung, heart, and kidney, as needed

All patients, whether or not they receive nitisinone, return to the Clinical Center for a 2-3 day follow-up admission every 4 months for a history and physical examination, blood tests, and two 24-hour urine collections. Every 12 months (12, 24 and 36 months after starting the study), patients also have repeat bone x-rays, spiral CT, kidney ultrasound, echocardiogram, and electrocardiogram. An Magnetic Resonance Imaging (MRI) of the brain is done at the end of the study.

Sixteen months after the end of the study enrollment period, the treated and non-treated groups are evaluated. If nitisinone has delayed the progression of joint disease in the treated group, the study continues and all patients receive the drug for the remainder of the study. If not, the study continues for another 20 months, at which time the study ends and the evaluation process is repeated.

Patients who develop symptoms such as corneal crystals, pain, or severe liver or nervous system toxicity may be taken off the study.

DETAILED DESCRIPTION:
Alkaptonuria is a rare metabolic disease in which homogentisic acid (HGA), an intermediary metabolite in tyrosine catabolism, accumulates due to deficiency of the enzyme homogentisic acid oxidase. Patients with alkaptonuria exhibit homogentisic aciduria and ochronosis, or dark pigmentation of various tissues due to binding of HGA and its oxidized metabolites. The ochronosis results in debilitating destruction of cartilage, arthritis, lumbosacral ankylosis, limitation of motion, and bone deterioration in later life. No effective therapy exists for alkaptonuria. However, a compound named 2-(2-nitro-4-trifluoromethylbenzoyl) - 1, 3-cyclohexanedione (nitisinone, NTBC, Orfadin) inhibits 4-hydroxyphenylpyruvate dioxygenase, the enzyme that produces HGA. Nitisinone, at doses of approximately 1 mg/kg/day, has proven safe and effective in tyrosinemia type I, which causes fatal liver disease in infants and children. Under protocol 97-HG-0201, we treated 9 alkaptonuria patients with nitisinone; for the 7 who received 1.05 mg twice daily, the HA fell from 4.0 plus or minus 1.8 g/24h to 0.2 plus or minus 0.2 g/24h (normal 0.028 plus or minus 0.015 g/24h, n=10). Plasma tyrosine levels rose from 67 plus or minus 18 micro M to 760 plus or minus 181 micro M. The current protocol (05-HG-0076) is a randomized, controlled clinical trial to determine if nitisinone (2 mg daily) is beneficial for the joint symptoms of alkaptonuira. Patients are examined at the NIH Clinical Research Center every 4 months for 3 years. Hip joint range of motion (ROM) serves as the primary outcome parameter, and nitisinone (Orfadin) is provided by Swedish Orphan International through an Investigational New Drug Application (IND), obtained by William A. Gahl. Forty patients (20 with nitisinone treatment and 20 untreated) have been enrolled for at least 16 months, and an interim analysis shows promising results. Serious adverse events in patients on nitisinone have included a death from myocardial infarction, keratopathy, and elevated liver function tests related to gallstones.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 30-80 years, either gender
* Diagnosis of alkaptonuria based upon urinary HGA excretion greater than 0.4 g/24h
* At least one hip joint remaining
* Some evidence of hip involvement, e.g., pain or decreased range of motion
* Ability to travel to the NIH Clinical Research Center for admissions
* Ability to consent
* Availability of local medical follow-up

EXCLUSION CRITERIA:

* Age less than 30 or greater than 80
* Non-alkaptonuria causes of ochronosis
* Bilateral hip joint replacement
* Keratopathy
* Contact lenses
* Uncontrolled glaucoma
* History of myocardial infarction
* History of emphysema or pulmonary insufficiency (Forced vital capacity less than 70%)
* Psychiatric illness or neurological disease that interferes with compliance or communication with health care personnel
* Current malignancy
* Open skin lesions
* Dietary habits or use of homeopathic therapies that interfere with tyrosine catabolism. The diet must be reasonably balanced, as determined by a dietician.
* Uncontrolled hypertension (blood pressure greater than 180 systolic or greater than 95 diastolic)
* History of extreme alcohol abuse or sever liver disease
* Liver greater than 3 cm below the right costal margin
* Electrocardiogram changes indicative of myocardial infarction, arrhythmia, tachycardia, bradycardia, left bundle branch block
* Chest radiographic abnormalities, including an infiltrate, mass, congestive heart failure, embolism, atelectasis
* Serum postassium less than 3. 0 mEq/L
* Serum creatinine greater than 2.0 mg/dL
* Serum glutamic-pyruvic transaminase (SGPT) greater than 41 U/L or Serum glutamic-oxaloacetic transaminase (SGOT) greater than 34 U/L
* Creatine kinase (CK) greater than 500 U/L
* Hemoglobin less than 10.0 g/dL
* Platelets less than 100 k/mm(3)
* White blood cells (WBCs) less than 3.0 k/microL
* Free thyroxine (T4) greater than 15 microg/dL
* T4 less than 4 microg/dL
* Erythrocyte sedimentation rate (ESR) greater than 100 mm/h
* Plasma tyrosine greater than 150 microM

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Introne WJ, Phornphutkul C, Bernardini I, McLaughlin K, Fitzpatrick D, Gahl WA. Exacerbation of the ochronosis of alkaptonuria due to renal insufficiency and improvement after renal transplantation. Mol Genet Metab. 2002 Sep-Oct;77(1-2):136-42. doi: 10.1016/s1096-7192(02)00121-x. PMID 12359141
- [Background] Phornphutkul C, Introne WJ, Perry MB, Bernardini I, Murphey MD, Fitzpatrick DL, Anderson PD, Huizing M, Anikster Y, Gerber LH, Gahl WA. Natural history of alkaptonuria. N Engl J Med. 2002 Dec 26;347(26):2111-21. doi: 10.1056/NEJMoa021736. PMID 12501223
- [Background] Janocha S, Wolz W, Srsen S, Srsnova K, Montagutelli X, Guenet JL, Grimm T, Kress W, Muller CR. The human gene for alkaptonuria (AKU) maps to chromosome 3q. Genomics. 1994 Jan 1;19(1):5-8. doi: 10.1006/geno.1994.1003. PMID 8188241
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-HG-0076.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at the NIH Clinical Center between April 2005 and March 2006.
Period: Overall Study
Arm/Group | Control | Nitisinone-treated
Started | 20 | 20
Completed | 17 | 16
Not Completed | 3 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Second hip replacement | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Nitisinone-treated | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 19 | 39
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (6.5) | 52.2 (7.9) | 51.7 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 15 | 12 | 27
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
Total Range of Motion (ROM) Worse Hip [Mean (Standard Deviation); unit: degrees] — The total (internal + external) range of motion (ROM) of the worse hip.
  degrees | 46.4 (16.1) | 39.0 (12.7) | 42.7 (14.8)
Schober's test [Mean (Standard Deviation); unit: cm] — Schober's test measures a patient's ability to flex his/her lower back. The examiner makes a mark at L5 (fifth lumbar vertebra) and places one finger 5 cm below and another finger 10 cm above this mark. The patient is asked to touch his/her toes. The examiner measures the increase in distance between the two fingers.
  cm | 11.42 (1.04) | 10.86 (0.73) | 11.14 (0.93)
Functional Reach Assessment [Mean (Standard Deviation); unit: cm] — Functional reach assessment measures the difference between the length of a person's outstretched arm and their maximal reach forward, while maintaining balance.
  cm | 10.22 (2.92) | 8.98 (3.10) | 9.60 (3.04)
Timed get up and go [Mean (Standard Deviation); unit: seconds] — In timed get up and go, the patient is asked to stand up from a standard chair and walk a distance of 3 meters, turn around and walk back to the chair and sit down. The examiner measures the time it takes for the patient to perform this series of tasks.
  seconds | 7.56 (1.40) | 9.70 (4.10) | 8.63 (3.21)
6 minute walk test [Mean (Standard Deviation); unit: ft] — The 6MWT measures the distance that a patient can quickly walk on a flat hard surface in a period of six minutes.
  ft | 1578 (205) | 1336 (369) | 1457 (319)

OUTCOME MEASURES:

1. Primary Outcome: Change in Total ROM Worse Hip
Description: Change from baseline in the total (external + internal) hip range of motion (ROM) in the worse hip at 36 months. The patient lies on exam table in the supine position. The patient flexes his/her hip and knee to 90 degrees. The examiner measures the patient's hip external rotation and hip internal rotation range of motion with a goniometer.
Time Frame: Measured at baseline and at 36 months
Population: Intention to treat.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control | Nitisinone-treated
Number analyzed (Participants) | 20 | 20
degrees | -9.1 (24.7) | 1.6 (21.8)

2. Secondary Outcome: Change in Schober's Test
Description: Change from baseline of Schober's test at 36 months. Schober's test measures a patient's ability to flex his/her lower back. The examiner makes a mark at L5 (fifth lumbar vertebra) and places one finger 5 cm below and another finger 10 cm above this mark. The patient is asked to touch his/her toes. The examiner measures the increase in distance between the two fingers.
Time Frame: Measured at baseline and at 36 months
Population: In the control group, two patients who dropped out for personal reasons were not included in this analysis, and in the treated group one patient who died was not included in this analysis.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Nitisinone-treated
Number analyzed (Participants) | 18 | 19
cm | -0.06 (1.33) | 0.12 (1.05)

3. Secondary Outcome: Change in Functional Reach Assessment
Description: Change from baseline of functional reach assessment at 36 months. Functional reach assessment measures the difference between the length of a person's outstretched arm and their maximal reach forward, while maintaining balance.
Time Frame: Measured at baseline and at 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Control | Nitisinone-treated
Number analyzed (Participants) | 18 | 19
cm | -1.21 (3.81) | -1.86 (3.59)

4. Secondary Outcome: Change in Timed Get up and go
Description: Change from baseline of timed get up and go at 36 months. In timed get up and go, the patient is asked to stand up from a standard chair and walk a distance of 3 meters, turn around and walk back to the chair and sit down. The examiner measures the time it takes for the patient to perform this series of tasks.
Time Frame: Measured at baseline and at 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Control | Nitisinone-treated
Number analyzed (Participants) | 18 | 19
seconds | -0.54 (1.84) | -1.33 (5.04)

5. Secondary Outcome: Change in 6 Minute Walk Test (6MWT)
Description: Change from baseline of the 6MWT at 36 months. The 6MWT measures the distance that a patient can quickly walk on a flat hard surface in a period of six minutes.
Time Frame: Measured at baseline and at 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ft
Arm/Group | Control | Nitisinone-treated
Number analyzed (Participants) | 18 | 19
ft | 22 (356) | 169 (591)

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Control | Nitisinone-treated
Serious Adverse Events (participants affected / at risk) | 0/20 | 6/20
Other Adverse Events (participants affected / at risk) | 10/20 | 10/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=20) | Nitisinone-treated (N=20)
atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
keratitis (Eye disorders) | 0 (0) | 1 (3) — corneal irritation due to tyrosine crystal deposition
bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1)
accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
liver enzyme elevation (Hepatobiliary disorders) | 0 (0) | 1 (1) — High elevations of alanine transaminase (ALT); ALT > 123 U/L.
muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
sarcoidosis (Immune system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Control (N=20) | Nitisinone-treated (N=20)
elevated liver enzymes (Hepatobiliary disorders) | 6 (8) | 6 (8) — Mild elevations in alanine transaminase (ALT); ALT between 41 and 100 U/L.
depression (Psychiatric disorders) | 2 (2) | 0 (0)
upper respiratory infection (Infections and infestations) | 5 (6) | 2 (2)
skin rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
sensorineural hearing loss (Ear and labyrinth disorders) | 0/0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
Small number of patients involved in study and several patients dropped out; primary outcome parameter selection possibly inappropriate because hip joint damage that is already present may be irreversible.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes